CLINICAL TRIAL: NCT06142617
Title: A Phase II Study of Pembrolizumab Plus Platinum and Pemetrexed as First Line Therapy in Advanced Non-squamous Non-small Cell Lung Cancer Patients With EGFR Exon 21 Point Mutation and Programmed Cell Death Ligand 1 Expression
Brief Title: A Prospective Study of Pembrolizumab Combining Chemotherapy in Advanced NSCLC Patients With EGFR Exon 21 Point Mutation.
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K4510
Record Dates: First submitted 2023-10-29; First posted 2023-11-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-10

CONDITIONS: Non Small Cell Lung Cancer; Immune Checkpoint Inhibitor; EGFR Exon 21 Mutation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab; Pemetrexed; Platinum; osimertinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental group (Experimental): Four cycles of platinum and pemetrexed in combination with pembrolizumab will be administered as first line therapy and up to 31 cycles pemetrexed and pembrolizumab maintenance therapy every 3 weeks. Osimertinib will be the sequential treatment strategy at progression until resistance develops.
  Interventions: Drug: Pembrolizumab, pemetrexed, platinum; Drug: Osimertinib

INTERVENTIONS:
Drug: Pembrolizumab, pemetrexed, platinum — Four cycles of platinum and pemetrexed in combination with pembrolizumab will be administered as first line therapy and up to 31 cycles pemetrexed and pembrolizumab maintenance therapy every 3 weeks.
  Other Names: Keytruda, pemetrexed, platinum
Drug: Osimertinib — Osimertinib will be the sequential treatment strategy at progression until resistance develops.

SUMMARY:
A phase II, single-arm, open-label study evaluating efficacy, safety and feasibility of combined chemotherapy and pembrolizumab as first line therapy and Osimertinib as second line therapy in advanced non squamous NSCLC adult patients with epidermal growth factor receptor (EGFR) exon 21 point mutation and programmed cell death receptor ligand 1 (PD-L1) positive.

DETAILED DESCRIPTION:
Four cycles of platinum and pemetrexed in combination with pembrolizumab will be administered as first line therapy and up to 31 cycles pemetrexed and pembrolizumab maintenance therapy every 3 weeks. Osimertinib will be the sequential treatment strategy at progression.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, ≥18 years old
2. Primary non-squamous non-small cell lung cancer(NSCLC) with stage IV (AJCC stage,8th Edition) confirmed by cytology or histology
3. Patients who have not used any anti-tumor therapy drugs such as targeted drugs, chemotherapy or immunotherapy and patients after surgery are acceptable
4. EGFR exon 21 point mutation confirmed by gene test of tissue or blood and PD-L1 (22C3) TPS≥1% confirmed by immunohistochemical method
5. At least one evaluable focus judged according to RECIST 1.1 standard
6. Eastern Cooperative Oncology Group performance score (PS) 0 or 1
7. Adequate blood function: absolute neutrophil count (ANC) ≥ 2 × 109 / L, platelet count ≥ 100 × 109 / L and hemoglobin 110 ≥ 9 g / dl. Adequate renal function: serum creatinine ≤ upper limit of normal value. Adequate liver function: total bilirubin ≤ upper limit of normal value(ULN); Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ upper limit of normal value (ULN); alkaline phosphatase ≤ upper limit of normal value (ULN)
8. Life expectancy is not less than 6 months
9. Male participants: Male participants must take effective contraception and do not donate sperm during the study and 180 days at least after the last dose
10. Female participants can not be pregnant, breastfeeding, and meet at least one of the following conditions:

    1. non-fertile women or
    2. agree to use effective contraception during treatment and 180 days at least after the last dose
    3. Fertile women must perform a serum or urine pregnancy test within 72 hours before the first dose and the results must be negative (minimum sensitivity 25 IU/L or human chorionic gonadotropin (HCG) equivalent unit)
11. Sign the informed consent form (the informed consent form needs to be approved by the independent ethics committee, and the informed consent of the patient should be obtained before starting any substantive trial procedure)

Exclusion Criteria:

1. patients who have active autoimmune disease which needs systemic treatment like disease relievers, corticosteroids, or immunosuppressants) in the last 2 years e. Alternative therapies ( such as thyroxine, insulin, and physiologic corticosteroid replacement therapy of adrenal or pituitary function insufficiency) are permitted)
2. History of pneumonia (non-infectious)/interstitial lung disease which require s steroid treatment or a current pneumonia/interstitial lung disease
3. Previously diagnosed immunodeficiency diseases, such as immunoglobulin deficiency, aplastic anemia
4. Known history of human immunodeficiency virus (HIV) infection
5. Patients who have hepatitis B (defined as hepatitis B virus (HBV) DNA > 1000 copy number) and hepatitis C virus (HCV) (defined as HCV RNA (+) infection
6. Known history of active tuberculosis infection
7. Patients who received live or attenuated vaccine within 30 days prior to the first study intervention and inactivated vaccines are allowed.
8. Patients who have other known malignancies within the past 1 year and needs treatment. Basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ that has undergone potentially curative treatment, and bladder carcinoma in situ are not included.
9. Patients who have symptomatic central nervous system metastases and/or meningitis
10. History of hypersensitivity ( ≥ Level 3) to pembrolizumab/pemetrexed/platinum/osimertinib and/or any of its excipients
11. Active infection that requires systemic treatment
12. Any medical condition that the investigator believes might do harm to the patient or not in the best interest of the patients such as poorly controlled diabetes, infection requiring treatment by injection, liver failure, mental illness or any disease, treatment, laboratory abnormality that might confuse the results or interfere with the participation of patients throughout the study.
13. Patients with mental illness or substance abuse which are confirmed to interfere with compliance with test requirements
14. Planed or currently pregnant or lactation during the study (from beginning of the screening visit to 180 days after the last dose of the experimental drug)
15. Patients who have undergone allogeneic tissue/solid organ transplantation
16. Patients who could not accept regular follow-up
17. Patients who are participating in or have used other investigational drugs or investigational equipment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2027-11-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
progression free survival 1 (PFS1) | up to 8 weeks
  the time length from enrollment to any of the following events: disease progression with first line therapy or death from any cause. Disease progression will be assessed according to RECIST 1.1

SECONDARY OUTCOMES:
progression free survival 2 (PFS2) | up to 8weeks
  the time length from enrollment to any of the following events: disease progression with Osimertinib or death from any cause. Disease progression will be assessed according to RECIST 1.1
Incidence of adverse events graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 | up to 8 weeks
  Evaluate adverse events of any cause, treatment-related adverse events, immune-mediated adverse events according to NCI-CTCAE V5.0
objective response rate (ORR) | up to 8 weeks
  Proportion of patients with Complete and Partial Responses to first-line therapy.
Life quality score | up to 8 weeks
  Evaluate life quality score according to Karnofsky performance status (KPS). On a scale of 10, higher scores indicate better health. A score of 0 is defined as death, on a 100-point scale, indicating normal physical fitness with no obvious symptoms and signs.

OTHER OUTCOMES:
Exploratory biomarker analysis | before treatment, at the time of disease progression on first-line therapy, and at the time of disease progression on second-line therapy.
  Blood samples will be collected from patients on three occasions: before treatment, at the time of disease progression on first-line therapy, and at the time of disease progression on second-line therapy. 15ml blood samples will be collected each time for PBMC assay. Tumor samples will be collected: 10 formalin-fixed, paraffin-embedded sections. Tumor samples will be subjected to genetic testing. Blood samples will be analyzed by flow cytometry.

CONTACTS AND LOCATIONS:
Overall Officials: Mengzhao Wang, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No
The result of the study and all the supporting information will be shared in the form of publishing article.